CLINICAL TRIAL: NCT01636739
Title: Special Drug Use Investigation for ROTARIX
Brief Title: Special Drug Use Investigation for ROTARIX®
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115927
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Infections, Rotavirus
Keywords: Intussusceptions; Special Drug Use Investigation; Rotavirus
MeSH Terms: conditions — Rotavirus Infections; Intussusception | interventions — RIX4414 vaccine; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rota Group: Subjects will receive Rotarix® as per routine practice
  Interventions: Biological: Oral Rotarix®; Other: Data collection

INTERVENTIONS:
Biological: Oral Rotarix® — 2 doses administered orally.
Other: Data collection — Additional information on intussusception will be collected through interview and by phone-contact.

SUMMARY:
This study aims to determine the incidence of intussusceptions (IS) (including suspected cases of intussusception) after vaccination with Oral Rotarix® under clinical practice, in Japan.

DETAILED DESCRIPTION:
This is non-interventional study conducted in one group received Oral Rotarix®.

ELIGIBILITY:
Inclusion Criteria:

* Infants who receive Rotarix for the first time to prevent rotavirus gastroenteritis, an indication of Rotarix, will be included in the investigation.

Exclusion Criteria:

* All infants included in the drug use investigation of Oral Rotarix will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants who receive Rotarix for the first time to prevent rotavirus gastroenteritis.
Sampling Method: Non-Probability Sample
Enrollment: 10982 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Determination of the incidence of IS | During the 31-day (Day 0 -Day 30) observation period after each vaccination
Determination of the incidence of IS | On the 1 year birthday of the subject

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline